CLINICAL TRIAL: NCT00150280
Title: A Prospective, Randomized, Double-Blind, Double-Dummy, Multi-Center Study Comparing Celecoxib and Ibuprofen Sr In The Management Of Acute Pain Post Orthopedic Or Gynecological Surgery
Brief Title: Compare Celecoxib and Ibuprofen Sr In The Management Of Acute Pain Post Orthopedic Or Gynecological Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191086
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Celecoxib

INTERVENTIONS:
Drug: celecoxib and ibuprofen SR

SUMMARY:
To validate the analgesic efficacy and safety of celecoxib compared with ibuprofen SR in the management of acute pain post orthopedic or gynecological surgery

ELIGIBILITY:
Inclusion Criteria:

* Undergone uncomplicated orthopedic surgery or abdominal gynecological surgery under epidural anesthesia
* Baseline pain intensity of more than 45 mm as measured by VAS and a severity of pain graded as moderate or severe on the categorical pain intensity scale

Exclusion Criteria:

* A previous history of intolerance or hypersensitivity to any NSAIDs, cyclooxygenase inhibitor, sulfonamides, or any analgesic, or to drugs with similar chemical structures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132
Dates: Start 2004-10; Study Completion 2005-07

PRIMARY OUTCOMES:
To validate the analgesic efficacy of celecoxib compared with ibuprofen SR in the management of acute pain post orthopedic or gynecological surgery

SECONDARY OUTCOMES:
To validate safety of celecoxib compared with ibuprofen SR in the management of acute pain post orthopedic or gynecological surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- China (3):
  - Pfizer Investigational Site, Shenyang, Liaoning
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai